CLINICAL TRIAL: NCT02589912
Title: Compassionate Use Arm - ABI541 Auditory Brainstem Implant for Neurofibromatosis Type 2 Patients With Deafness
Brief Title: Compassionate Use Arm - ABI541 ABI for 10 NF2 Patients
Status: No longer available | Type: Expanded Access
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Dr. Daniel Lee, Attending Physician, Massachusetts Eye and Ear Infirmary
Other Study IDs: 15-113H
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Neurofibromatosis Type 2; Severe Profound Sensorineural Hearing Loss
MeSH Terms: conditions — Neurofibromatosis 2

INTERVENTIONS:
Device: Nucleus Profile ABI541 Auditory Brainstem Implant

SUMMARY:
The Nucleus 24 Auditory Brainstem Implant (ABI) is the only FDA approved device for restoration of meaningful hearing in Neurofibromatosis Type 2 (NF2) patients. This device has been discontinued, meaning that there is no commercially approved device currently available. The replacement model, the ABI541 (an unapproved device), is being investigated in ongoing clinical trials. A compassionate use arm of a clinical trial allows patients with NF2 to be implanted with this new ABI.

DETAILED DESCRIPTION:
Currently, the Nucleus 24 (ABI24M) Auditory Brainstem Implant (ABI) is approved for use in individuals 12 years of age or older who have been diagnosed with Neurofibromatosis Type 2 (NF2). Implantation may occur during first or second side tumor removal or in patients with previously removed vestibular schwannomas bilaterally. As the ABI24M is now obsolete, there is currently no commercially approved device available to restore useful hearing in patients. While the manufacturer of the device is pursuing commercial approval of the ABI541, it is anticipated that it may be several months or years before final approval. However, it is preferable to place the device at the time of tumor removal while the patient has an open craniotomy site, thereby avoiding a second surgery and its associated risks solely for the purpose device implantation. In addition, placement of an ABI at the time of tumor removal optimizes auditory rehabilitation, providing critical auditory sensations that may more effectively maintain auditory pathways. The FDA approved a compassionate use arm for an ongoing clinical trial to permit implantation of the ABI541 in up to 10 NF2 patients.

Patients will undergo pre-operative evaluation for ABI surgery. Those who are appropriate for surgery will undergo a procedure for implantation of the ABI541. As per manufacturer protocol, the parameters of the ABI541 including adjustment of electrode sensitivities and activation of specific electrodes will be completed at each follow-up visit post-operatively. This process involves adjustment of device parameters by a trained audiologist who subsequently administers audiologic tests to confirm optimal activation of the ABI541.

All audiologic testing and assessments represent the standard of care. These post-operative follow-up appointments will occur at 4-12 weeks, three, six, and twelve months, and biannually thereafter. Timing of these appointments may vary by as much as four weeks prior to or after the planned follow-up date (e.g. between 2-4 months for the 3 month follow-up). Unscheduled visits will be taken in the Otology clinic as needed to address any concerns patients may have regarding the use of their Nucleus ABI541.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Neurofibromatosis Type 2;
* Age of 12 years or older
* Will be anticipated to be completely deaf as a result of bilateral neurofibromas of the auditory nerve, and/or their surgical removal.

Exclusion Criteria:

* Contraindications to surgery or general anesthesia
* Intractable seizures or progressive, deteriorating neurological disorder
* Unable to participate in behavioral testing and mapping with ABI
* Unrealistic expectations on the part of the subject/family regarding possible benefits, risks, and limitations that are inherent to the procedure and prosthetic device

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States